CLINICAL TRIAL: NCT02656875
Title: A Phase 3, Open-label Study to Evaluate the Safety of TRV130 in Patients With Acute Pain for Which Parenteral Opioid Therapy is Warranted
Brief Title: A Open-label Study to Evaluate the Safety of TRV130 in Patients With Acute Pain
Acronym: ATHENA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP130-3003
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRV130 (Experimental): For clinician-administered bolus dosing, TRV130 initial dose is administered and supplemental dosing is available, if clinically indicated. Subsequent doses may be administered every 1 to 3 hours as needed.
  For PCA dosing, the TRV130 regimen consists of a loading dose, a demand dose, and a lockout interval.
  Interventions: Drug: TRV130

INTERVENTIONS:
Drug: TRV130
  Other Names: oliceridine

SUMMARY:
Patients with moderate to severe pain caused by medical conditions or surgery, who require IV opioid therapy may be enrolled in this open label safety study. Patients will be treated with TRV130 by IV bolus, PCA (patient-controlled analgesia) administration, or both, as determined by the investigator, for a duration not to exceed 14 days.

DETAILED DESCRIPTION:
The duration of treatment for each patient will be determined by the clinical need for parenteral opioid therapy. Eligible patients with moderate to severe pain caused by medical conditions or surgery, who require IV opioid therapy may be enrolled in this open label safety study. Patients will be treated with TRV130 by IV bolus, PCA administration, or both, as determined by the investigator, for a duration not to exceed 14 days. The duration of treatment for each patient will be determined by the clinical need for parenteral opioid therapy. A follow-up assessment will take place 2-3 days after the completion of the treatment phase.

ELIGIBILITY:
Inclusion Criteria include:

* Moderate to severe acute pain for which parenteral opioid therapy is warranted
* Able to understand and comply with the procedures and study requirements, and to provide written informed consent before any study procedure.

Exclusion Criteria include:

* Clinically significant medical, surgical, postsurgical, psychiatric or substance abuse condition or history of such condition that would confound the interpretation of safety, tolerability, or efficacy data in the study.
* Hemodynamic instability or respiratory insufficiency.
* Advanced cancer in palliative or end-of-life care.
* Another current painful condition (other than acute pain for which parenteral opioid therapy is warranted) that would confound the interpretation of safety, tolerability, or efficacy data in the study.
* Clinically significant, immune-mediated hypersensitivity reaction to opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, MD, Study Chair — Trevena Inc.
Locations (9):
- United States (9):
  - Recruiting, Mobile, Alabama
  - Recruiting, Pasadena, California
  - Recruiting, Miami, Florida
  - Recruiting, Shreveport, Louisiana
  - Recruiting, Jackson, Mississippi
  - Staten Island, New York
  - Recruiting, State College, Pennsylvania
  - Houston, Texas
  - Recruiting, Murray, Utah

REFERENCES:
- [Derived] Bergese SD, Brzezinski M, Hammer GB, Beard TL, Pan PH, Mace SE, Berkowitz RD, Cochrane K, Wase L, Minkowitz HS, Habib AS. ATHENA: A Phase 3, Open-Label Study Of The Safety And Effectiveness Of Oliceridine (TRV130), A G-Protein Selective Agonist At The micro-Opioid Receptor, In Patients With Moderate To Severe Acute Pain Requiring Parenteral Opioid Therapy. J Pain Res. 2019 Nov 14;12:3113-3126. doi: 10.2147/JPR.S217563. eCollection 2019. PMID 31814753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRV130
Started | 768
Completed | 698
Not Completed | 70

BASELINE CHARACTERISTICS:
Groups:
- TRV130: For clinician-administered bolus dosing, TRV130 initial dose is administered and supplemental dosing is available, if clinically indicated. Subsequent doses may be administered every 1 to 3 hours as needed.
  For PCA dosing, the TRV130 regimen consists of a loading dose, a demand dose, and a lockout interval.
  TRV130
Arm/Group | TRV130
Number analyzed (Participants) | 768
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 521
  >=65 years | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (16.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 498
  Male | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 596
  Black or African American | 137
  Asian | 13
  American Indian or Alaska Native | 5
  Native Hawaiian or Other Pacific Islander | 1
  Other | 14
  Missing Race | 2
  Hispanic or Latino | 61
  Not Hispanic or Latino | 704
  Missing Ethnicity | 3
Region of Enrollment [Number; unit: participants]
  United States | 768

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experienced a Treatment-emergent Adverse Event
Time Frame: From first dose through 3 days after last dose, approximately 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | TRV130
Number analyzed (Participants) | 768
Participants | 490

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dose through the follow-up visit, which occurred up to 3 days after last dose (approximately 4 days total).
Description: Adverse events were collected from time of first dose through the follow-up visit, which occurred up to 3 days after last dose (approximately 4 days total). Serious Adverse Events were collected from informed consent through 7 days following last dose.
Arm/Group | TRV130
All-Cause Mortality (participants affected / at risk) | 0/768
Serious Adverse Events (participants affected / at risk) | 26/768
Other Adverse Events (participants affected / at risk) | 403/768
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRV130 (N=768)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Graft Infection (Infections and infestations) | 1 (1)
Pelvic Abscess (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Anemia Postoperative (Injury, poisoning and procedural complications) | 1 (1)
Postprocedural Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Postprocedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Breast Hematoma (Reproductive system and breast disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRV130 (N=768)
Nausea (Gastrointestinal disorders) | 239
Constipation (Gastrointestinal disorders) | 84
Vomiting (Gastrointestinal disorders) | 80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02656875/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT02656875/SAP_001.pdf